CLINICAL TRIAL: NCT02324088
Title: Phase III Trial Assessing the Interest of a Maintenance Chemotherapy Combining Docetaxel (Taxotere) 5-FU After Induction Treatment by Aintensive Chemotherapy for Inflammatory Breast Cancers
Brief Title: Interest of Maintenance Chemotherapy After Induction Treatment for Inflammatory Breast Cancer
Acronym: PEGASE07
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEGASE 7/0002
Record Dates: First submitted 2014-12-14; First posted 2014-12-24 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Inflammatory Breast Cancer
MeSH Terms: conditions — Inflammatory Breast Neoplasms | interventions — Docetaxel; Cyclophosphamide; Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): 4 cycles of high-dose EC (E150 mg/m² and C 4000 mg/m² every 3 weeks) then mastectomy with axillary lymph node dissection and radiotherapy
  Interventions: Drug: Cyclophosphamide; Drug: Epirubicin
- Arm B (Experimental): 4 cycles of high-dose EC (E150 mg/m² and C 4000 mg/m² every 3 weeks) then mastectomy with axillary lymph node dissection and radiotherapy followed by 4 cycles of D-5FU (D 85 mg/m², day 1 and 5FU 2500 mg/m²/day continuous infusion, days 1-5 every 3 weeks)
  Interventions: Drug: Docetaxel; Drug: Cyclophosphamide; Drug: Epirubicin

INTERVENTIONS:
Drug: Docetaxel
  Arms: Arm B
Drug: Cyclophosphamide
Drug: Epirubicin

SUMMARY:
To evaluate the benefit of adding docetaxel-5 fluorouracile (D-5FU) regimen after pre-operative epirubicin-cyclophosphamide (EC) and loco-regional treatment in inflammatory breast cancer (IBC).

ELIGIBILITY:
Inclusion Criteria:

* histologically proven breast cancer
* inflammatory breast cancer
* no metastatic site
* age > or = 18 and < or = 60
* OMS score: 0, 1, 2
* life expectancy > or = 3 months
* Normal (isotopic or ultrasonography) left ventricular ejection fraction
* Normal haematological, liver, and kidney functions
* patients who gave their written informed consent.

Exclusion Criteria:

* non inflammatory breast tumour with a cutaneous permeation nodule
* presence of a metastatic site
* medical history of a cancerous tumour except for carcinoma in situ of the uterine cervix, a basal cell skin cancer, or a breast carcinoma on the contralateral side
* patients having already had a chemotherapy, a radiotherapy, or an hormone therapy for this breast tumour
* medical history of congestive heart failure even medically controlled
* medical history of myocardial infarction during the 6 months before the inclusion in the study
* active infection or other severe underlying pathology which could possibly prevent the patient from receiving treatments
* administration of another chemotherapy during the study
* pregnant or breast feeding patients (the patients of childbearing age must be placed under efficient contraception)
* patients whose social or psychological state does not allow to consider a correct adherence to the treatment and to the required medical follow-up
* WHO score 3,4
* unbalanced diabetes
* polysorbate 80 allergy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 174 (Actual)
Dates: Start 2000-10; Primary Completion 2012-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
disease-free survival rate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Viens, MD, Principal Investigator — Institut Paoli Calmette Marseille

IPD SHARING:
Plan to Share IPD: Yes
Unicancer will share de-identified individual data that underlie the results reported. A decision concerning the sharing of other study documents, including protocol and statistical analysis plan will be examined upon request.
Time Frame: Unicancer will consider access to study data upon written detailed request sent to Unicancer, from 6 months until 5 years after publication of summary data.
Access Criteria: The data shared will be limit to that required for independent mandated verification of the published results, the applicant will need authorization from Unicancer for personal access, and data will only be transferred after signing of a data access agreement.

REFERENCES:
- [Result] Goncalves A, Pierga JY, Ferrero JM, Mouret-Reynier MA, Bachelot T, Delva R, Fabbro M, Lerebours F, Lotz JP, Linassier C, Dohollou N, Eymard JC, Leduc B, Lemonnier J, Martin AL, Boher JM, Viens P, Roche H. UNICANCER-PEGASE 07 study: a randomized phase III trial evaluating postoperative docetaxel-5FU regimen after neoadjuvant dose-intense chemotherapy for treatment of inflammatory breast cancer. Ann Oncol. 2015 Aug;26(8):1692-7. doi: 10.1093/annonc/mdv216. Epub 2015 May 5. PMID 25943350